CLINICAL TRIAL: NCT03745690
Title: Phase 1B/2, Open-Label Study Evaluating Safety and Efficacy of Enhanced Permeability and Retention Effect for Near-Infrared Image Guided Surgical Resection of Head and Neck Cancers With Indocyanine Green
Brief Title: Near-Infrared Image Guided Surgical Resection With Indocyanine Green in Treating Patients With Head and Neck Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: no enrollment
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-000168; NCI-2018-02094 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18-000168 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Head and Neck Carcinoma
MeSH Terms: interventions — Surgery, Computer-Assisted; Indocyanine Green; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (near-infrared image guided surgical resection) (Experimental): Patients receive indocyanine green IV on day 0 and undergo near-infrared image guided surgical resection on day 1.
  Interventions: Procedure: Image-Guided Surgery; Drug: Indocyanine Green Drug

INTERVENTIONS:
Procedure: Image-Guided Surgery — Undergo near-infrared image guided surgical resection
Drug: Indocyanine Green Drug — Given IV
  Other Names: IC-GREEN; ICG Drug in solution

SUMMARY:
This phase Ib/II trial studies the side effects of near-infrared image guided surgical resection with indocyanine green in treating patients with head and neck cancer. Near-infrared image guided surgical resection with indocyanine green may make it easier to find and remove tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety profile of high-dose optical dye, indocyanine green, in head and neck cancer surgical patients.

SECONDARY OBJECTIVES:

I. Determine the efficacy of high-dose indocyanine green to identify cancer compared to surrounding normal tissue (tumor to background ratio; TBR) in head and neck cancer resections.

OUTLINE:

Patients receive indocyanine green intravenously (IV) on day 0 and undergo near-infrared image guided surgical resection on day 1.

After completion of study treatment, patients are followed up for 14-30 days.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of a head and neck cancer diagnosis as evidenced by tissue biopsy.
* Patients diagnosed with any T stage, any subsite within the head and neck that are scheduled to undergo surgical resection. Patients with recurrent disease or a new primary will be allowed.
* Planned standard of care surgery with curative intent for squamous cell carcinoma.
* Have life expectancy of more than 12 weeks.
* Karnofsky performance status of at least 70% or Eastern Cooperative Oncology Group (ECOG)/Zubrod level 1.
* Hemoglobin >= 9 gm/dL.
* White blood cell count > 3000/mm^3.
* Platelet count >= 100,000/mm^3.
* Serum creatinine =< 1.5 mg/dL.
* Liver enzymes (aspartate aminotransferase [AST], alanine aminotransferase [ALT], and total bilirubin) =< 1.5 times the upper reference range.
* Written informed consent (and assent when applicable) obtained from subject or subject?s legal representative and ability for subject to comply with the requirements of the study.
* Agree to not have radioactive iodine uptake studies done within 1 week of indocyanine green.

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
* Allergy to iodine or iodinated materials.
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data.
* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-06-08 (Estimated); Study Completion 2021-06-08 (Estimated)

PRIMARY OUTCOMES:
Safety related by type, incidence, severity, seriousness, and study treatment relatedness of adverse events | Up to 30 days
  Adverse events will be tabulated by treatment group and will include the number of patients for whom the event occurred, the rate of occurrence, and the severity and relationship to study drug.

SECONDARY OUTCOMES:
Successful tumor fluorescence imaging data gathered for all patients included in the study | Up to 30 days
  The effect of indocyanine green will be assessed by changes in tumor-to-background ratio (TBR). Tumor to background (TBR) data will be generated from still images collected throughout the procedure as previously described (Heath, Deep et al.). The presence of fluorescence in normal surrounding tissue will be correlated with fluorescence within the tumor mass. The linear relationship between fluorescence and tumor size will be computed as Spearman?s correlation coefficient. Continuous variable means (e.g., fluorescence intensity) will be compared to histological quantification of tumor as measured by the greatest dimension identified on the histopathological assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Abie Mendelsohn, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States